CLINICAL TRIAL: NCT02895854
Title: LDR Brachytherapy Versus Hypofractionated SBRT for Low and Intermediate Risk Prostate Cancer Patients
Brief Title: LDR Brachytherapy Versus SBRT for Low and Intermediate Risk Prostate Cancer Patients
Acronym: BRAVEROBO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUH5654155
Record Dates: First submitted 2013-09-09; First posted 2016-09-12 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer
Keywords: Low risk prostate cancer; Intermediate risk prostate cancer; Low dose-rate brachytherapy; Hypofractionated; Robotic external beam radiation; Quality of life
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LDR-brachytherapy with I125 seeds (Active Comparator): Low-dose rate-brachytherapy with I125 permanent seeds in prostate cancer.
  Interventions: Radiation: LDR-brachytherapy with I125 seeds
- Hypofractionated RT 5 x 7,25 Gy (Active Comparator): Hypofractionated stereotactic radiotherapy 5 x 7,25 Gy delivered every second day in prostate cancer.
  Interventions: Radiation: Hypofractionated RT 5 x 7,25 Gy

INTERVENTIONS:
Radiation: Hypofractionated RT 5 x 7,25 Gy
  Arms: Hypofractionated RT 5 x 7,25 Gy
Radiation: LDR-brachytherapy with I125 seeds
  Arms: LDR-brachytherapy with I125 seeds

SUMMARY:
The aim of this trial is to find out if there are any differences in the profiles of acute and late adverse effects among men with low and intermediate risk prostate cancer treated either with low dose-rate brachytherapy or hypofractionated external radiotherapy (CyberKnife). Also the prostate specific antigen (PSA) responses and cost utility of each treatment will be analysed.

DETAILED DESCRIPTION:
Prostate cancer (PC) is the most common solid malignancy among the men in the Western world. The classification to low, intermediate and high risk groups is determined by the PSA, Gleason score and clinical TNM status at the moment of diagnosis. There are several treatment options available for patients with low and intermediate risk PC and generally their prognosis is good. The men live long after their radical treatments and they have to live with the possible adverse effects caused by the treatment.

In this prospective, randomised clinical trial we are comparing two radiotherapy modalities to find out if there are differences in the acute and late adverse effects among men treated either by low dose-rate (LDR) brachytherapy or hypofractionated external radiotherapy. Also the PSA-responses and cost utilities will be analysed. The number of patients recruited for the study is 60 and the patients will be randomised 1:1 to each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* biopsy proven adenocarcinoma of the prostate
* Gleason score ≤ 3+4
* clinical and radiological TNM T1c-2c, N0-X, M0-X, PSA ≤ 20ng/ml and WHO 0-2
* low or intermediate risk prostate cancer according to National Comprehensive Cancer Network (NCCN) classification

Exclusion Criteria:

* clinical TNM ≥ T3
* Gleason score ≥ 4+3
* high risk prostate cancer according to NCCN classification
* history of cancer (other than PC) during the past 5 years (excluding basalioma and squamocellular carcinoma of the skin)
* previous pelvic radiotherapy
* previous active treatments of prostate cancer (active surveillance allowed)
* bilateral hip prothesis or other implant impedes pelvic TT or MRI imaging
* clopidogrel medication
* poor co-operation
* life expectancy < 5 yrs

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-01-08 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in acute adverse effects | 6 months
  questionnaires

SECONDARY OUTCOMES:
Time to PSA response | 6 months
Time to PSA nadir | 2 years
Biological progression free survival (bPFS) | 3 years

OTHER OUTCOMES:
Cost utility | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kristiina Vuolukka, MD, Principal Investigator — Cancer Center, KUH
Locations (1):
- Kuopio University Hospital, Kuopio, Finland